CLINICAL TRIAL: NCT00064285
Title: Phase I Study Of Flavopiridol In Combination With Imatinib Mesylate (STI571, Gleevec) In Bcr/Abl+ Hematological Malignancies
Brief Title: Flavopiridol and Imatinib Mesylate in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: National Cancer Institute
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000310175; U01CA062502 (NIH); MCV-NCI-6013; MCV-VCU-1902; NCI-6013; CWRU-030323
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2010-05-03 (Estimated); Status verified 2010-04

CONDITIONS: Leukemia
Keywords: chronic phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; recurrent adult acute myeloid leukemia; untreated adult acute myeloid leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; recurrent adult acute lymphoblastic leukemia; untreated adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Blast Crisis; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Congenital Abnormalities | interventions — alvocidib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: alvocidib
Drug: imatinib mesylate

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth. Drugs used in chemotherapy such as flavopiridol use different ways to stop cancer cells from dividing so they stop growing or die. Combining imatinib mesylate with flavopiridol may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of flavopiridol and imatinib mesylate in treating patients with hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and recommended phase II dose of flavopiridol and imatinib mesylate in patients with Bcr/Abl+ hematological malignancies.
* Determine the toxic effects of this regimen in these patients.
* Determine the disease-related effects of this regimen in these patients.
* Determine the pharmacokinetics and pharmacodynamics of this regimen in these patients.
* Correlate response to this regimen with mechanisms of imatinib mesylate resistance in patients previously treated with imatinib mesylate.

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to percentage of blasts in the peripheral blood and bone marrow (less than 15% vs at least 15%) and recent myelosupressive treatment (no vs yes).

Patients receive oral imatinib mesylate daily and flavopiridol IV over 1 hour on days 2, 9, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of imatinib mesylate and flavopiridol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 6-80 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Chronic or accelerated phase chronic myelogenous leukemia (CML) with 1 of the following:

    * Hematologic progression during prior imatinib mesylate treatment
    * Less than a complete hematologic response after at least 3 months of prior imatinib mesylate treatment
    * Less than a major cytogenetic response after at least 6 months of imatinib mesylate treatment (cytogenetic response documented by karyotype or fluorescence in situ hybridization [FISH])
  * Blastic phase CML*
  * Acute lymphoblastic leukemia*
  * Acute myeloid leukemia* NOTE: *Patients may be enrolled at presentation, in remission, or upon relapse
* Bcr/Abl+ in bone marrow confirmed by karyotype or FISH
* No known CNS malignancy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 2.5 times ULN (5 times ULN if hepatic involvement suspected [stratum 2 only])

Renal

* Creatinine no greater than 2 times ULN

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 3 months after study participation
* No prior allergic reaction attributed to compounds of similar chemical or biological composition to study agents
* No other concurrent uncontrolled medical illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent filgrastim (G-CSF), sargramostim (GM-CSF), or interleukin-2 during the first course of study therapy unless clinically indicated for management of febrile neutropenia or thrombocytopenia
* Concurrent epoetin alfa allowed if started before study entry and it remains clinically appropriate

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* See Disease Characteristics
* Recovered from all prior therapy
* No other concurrent investigational or anticancer agents
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2003-06

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grant, MD, Study Chair — Massey Cancer Center
Locations (4):
- United States (4):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Ireland Cancer Center at University Hospitals of Cleveland and Case Western Reserve University, Cleveland, Ohio
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia